CLINICAL TRIAL: NCT05222516
Title: A Randomised, Double-Blind, Placebo-controlled, 32-week, Phase IIa Trial to Investigate the Efficacy of OM-85 Versus Matched Placebo in Reducing Disease Severity Children Aged 3 to 24 Months With Early Clinical Diagnosis of Moderate Atopic Dermatitis
Brief Title: Immunomodulation by OM-85 (Broncho-Vaxom) in Early AD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recommendation of DSMB (futility of Endpoints)
Sponsor: OM Pharma SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BV-2021/06
Record Dates: First submitted 2021-12-22; First posted 2022-02-03 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-04

CONDITIONS: Atopic Dermatitis
Keywords: Moderate, Children
MeSH Terms: conditions — Dermatitis, Atopic; Lymphoma, Follicular | interventions — Broncho-Vaxom

STUDY DESIGN:
Intervention Model Description: OM-85 vs. placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Multicenter, randomized, double blind, placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OM-85 (Experimental): Daily administration of OM-85 (Broncho-Vaxom) 3.5 mg capsules
  Interventions: Drug: Broncho-Vaxom
- Placebo (Placebo Comparator): Daily administration of Placebo capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Broncho-Vaxom — Daily administration of Broncho-Vaxom 3.5mg capsules
  Other Names: OM-85
  Arms: OM-85
Drug: Placebo — Daily administration of Placebo capsules
  Arms: Placebo

SUMMARY:
Clinical data suggest that treatment with OM-85, by inducing an early contact with bacterial extracts, could modulate the immunity of children with Atopic Dermatitis, and thus play an active role in the treatment of Atopic Dermatitis.

The present trial will investigate the influence of administration of OM-85 in the paediatric population younger than 24 months with moderate atopic dermatitis.

The efficacy and safety of OM-85 will be evaluated in children aged 3 to 24 months old with moderate Atopic Dermatitis who may benefit from treatment with OM-85. The placebo treatment period will serve as a reference and has been added to establish efficacy and safety.

DETAILED DESCRIPTION:
In this study, the efficacy of OM-85 versus matched placebo in children with moderate AD (Atopic Dermatitis) in reducing disease severity shall be evaluated.

Clinical data suggest that treatment with OM-85, by inducing an early contact with bacterial extracts, could modulate the immunity of children with AD, and thus play an active role in the treatment of AD.

This will be a multicenter, randomised, double-blind, placebo-controlled exploratory phase IIa trial to assess the efficacy and safety of daily oral administration of OM-85 or matched placebo in children aged 3 to 24 months for 24 weeks.

A total of 142 children with AD as defined by Hanifin and Rajka criteria and with moderate disease severity (EASI 7.1 - 21.0) at Screening will be enrolled into this trial in approximately 15 sites in Germany and potentially one additional European country. All screened subjects will receive a unique subject ID (Identification) number.

Eligible subjects will be randomized at 1:1 ratio, stratified by age (≤12 months vs. >12 months) and disease severity (EASI <16 vs. ≥16) to one of the two treatments. They will receive either OM-85 or placebo for a 24-week treatment period followed by an observational period of 8 weeks without investigational medicinal products (IMP).

The placebo will serve as reference in evaluating efficacy and safety of OM-85. The double blind, randomized trial design is selected to avoid bias concerning evaluation of the drug effects, including safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Children of either gender, aged 3 to 24 months
* Patients with a clinically confirmed diagnosis of AD (according to Hanifin and Rajka) of moderate severity (EASI 7.1 - 21.0) and lesions covering up to 30% of the body either assessed by Investigator at the Screening/Baseline visit or recently (<4 weeks prior to Screening/Baseline visit) documented by Investigator and pre-treated with TCS (within last 4 weeks prior to Screening/Baseline visit).
* Atopic Dermatitis onset no longer than 12 months before Screening
* Legally acceptable representatives (i.e. parent(s) or guardians) of subject according to local regulations have provided the appropriate written informed consent. Written informed consent must be provided before any study specific procedures are performed including Screening procedures.

Exclusion Criteria:

* Any diseases that may be considered as the differential diagnosis of atopic dermatitis, and notably skin infections and infestations (e.g. scabies), other inflammatory skin conditions, dermatological malignancies, dermatological genetic diseases such as immunodeficiency conditions, and nutritional disorders with cutaneous manifestations and drug eruptions.
* Specifically, any inflammatory skin conditions that are considered during the differential diagnosis of atopic dermatitis: allergic contact dermatitis, dermatographism, psoriasis, pityriasis alba.
* Any chronic diseases (other than wheezing and asthmatic bronchitis) that require the administration of systemic corticosteroids (e.g., eosinophilic esophagitis) or immunosuppressant agents.
* Significant medical condition(s), which, in the Investigator's opinion, are anticipated to require major surgery during the study, or any other type of disorder that might involve an increased risk to the subject, could interfere with study assessments or outcomes, or the ability of parents to comply with the study procedures (e.g. eDiary).
* Infants and children with known allergy or previous intolerance/sensitivity to any of the trial treatments (IMP, AxMP or standardized emollient) to be administered.
* Use of systemic drugs interfering with the immune system (e.g. corticosteroids, immunosuppressants) within 30 days before Baseline (with exception of routine vaccinations)
* Previous or ongoing treatment with other bacterial lysates and/or probiotics within 30 days before Baseline
* Use of systemic antibiotics within 30 days before Baseline
* Participation in any other investigational trial on a medical device or medicinal product <30 days prior to Baseline or any previous participation in a study involving bacterial lysates and/or probiotics, or current treatment with other investigational agent(s)
* Any major surgery within the last 3 months prior to Baseline, that in the opinion of the Investigator, would not allow safe completion of the clinical study.
* Subject's families expected to relocate out of study area during the duration of the study.
* Other household members have previously been randomised in this clinical study.
* Previous participation to this study.
* Close affiliation of subject or parents with the investigational site; e.g. a close relative of the Investigator, dependent person (e.g. employee or student of the investigational site)

Ages: 3 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2023-07-13 (Actual)

PRIMARY OUTCOMES:
Disease severity | 16 weeks
  - Weekly area under the curve (AUC) of the EASI score from baseline to the latest evaluable assessment before or on week 16 visit, use of rescue medication, loss to follow-up or withdrawal of consent, whichever occurs first.
Disease severity | 24 weeks
  - Weekly area under the curve (AUC) of the EASI score from baseline to the latest evaluable assessment before or on week 24 visit, use of rescue medication, loss to follow-up or withdrawal of consent, whichever occurs first.

SECONDARY OUTCOMES:
Frequency of flares | 32 Weeks
  - Time to new AD flare, defined as ≥ 50% worsening of Baseline EASI score or EASI score of > 21.0 (severe AD) from Baseline to end of the treatment period and the observational period.
Reduction of flares | 24 Weeks
  - Percentage of patients free of flares from Baseline to the end of treatment period
Change of flares | 24 Weeks
  - Difference in free of flares days between treatment groups (placebo vs. verum) from Baseline to the end of treatment period
Number of flares | 32 Weeks
  - Number of new AD flares during the induction and maintenance period and during the whole treatment and observational period
Disease severity treatment period | 24 weeks
  - Weekly AUC of the EASI score from Baseline to the end the treatment period
Disease severity observational | 32 weeks
  - Weekly AUC of the EASI score from Baseline to the end of the observational period
EASI change | 32 weeks
  - EASI score change during the induction and maintenance period and during the whole treatment period and the observational period.
Scorad change | 32 weeks
  SCORAD score change during the induction and maintenance period and during the whole treatment period and the observational period
vIGA-AD change | 32 weeks
  - vIGA-AD (Validated Investigator Global Assessment in Atopic Dermatitis) score change during the induction and maintenance period and during the whole treatment period and the observational period
ADCT change | 32 weeks
  - ADCT score change during the induction and maintenance period and during the whole treatment period and the observational period
Co-medication use per patient | 32 weeks
  - Number and duration in days of TCS (Topical Corticosteroids) treatments for acute flares during the induction and maintenance period and during the whole treatment period and the observational period
Skin infections and systemic treatment | 32 weeks
  - Incidence of skin infections requiring systemic treatment and antibiotics during the induction and maintenance period and during the whole treatment period and the observational period
Respiratory tract infections | 32 weeks
  - Number of respiratory tract infections and wheezing episodes during the induction and maintenance period and during the whole treatment period and the observational period

OTHER OUTCOMES:
Immunomodulatory effects of OM-85 | 32 weeks
  - Change of gut microbiome from Baseline to the end of the treatment period and to the observational period.
Skin/gut microbiome | 32 weeks
  - Change of skin microbiome during the induction and maintenance period and during the whole treatment period and the observational period, incl. S. Aureus infections.
Correlation of microbiomes and outcomes | 32 weeks
  - Potential correlations between gut microbiome data and primary and/or secondary outcomes (e.g., EASI, SCORAD, vIGA-AD).
Correlation of gut microbiome and skin microbiome | 32 weeks
  - Potential correlations between gut microbiome data and skin microbiome and primary and/or secondary outcomes (e.g. EASI, Scorad, vIGA-AD) data (using diversity measures for the skin microbiome)
Allergic sensitisation IgE | 32 weeks
  - Optional: Change of total IgE ( Immunoglobulin E) and specific IgEs from Baseline to the end of the treatment period and the observational period
Allergic sensitisation biomarkers | 32 weeks
  - Optional: Change in expression of disease biomarkers in blood from Baseline to the end of the treatment period and the observational period.
OM-85 treatment-emergent adverse events and treatment-emergent serious adverse events | 32 weeks
  - Incidence of treatment-emergent adverse events and treatment-emergent serious adverse events from Baseline to the end of the observational period
Skin/gut microbiome | 32 weeks
  Potential correlations between skin microbiome data and primary and/or secondary outcomes (e.g., EASI, SCORAD, vIGA-AD)

CONTACTS AND LOCATIONS:
Overall Officials: Franziska Rueff, Professor, Principal Investigator — Universitätsklinikum München
Locations (28):
- France (6):
  - Centre d'investigation clinique GHE, Bron
  - CHU de Cote de Nacre, Centre de Recherche Clinique Pediatric, Caen
  - Hopital Hotel Dieu, Nantes
  - CHU de Nice, Nice
  - CHU de Poitiers, L'unité de Dermatologie, Poitiers
  - Mediopole Hopital Mutualiste, Villeurbanne
- Germany (17):
  - ISA - Interdisciplinary Study Association GmbH, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Elbe Klinikum Buxtehude, Buxtehude
  - Universitätsklinikum Dresden, Dresden
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - MENSINGDERMA research GmbH, Hamburg
  - Kinderhautarztpraxis Dr. Marc Pleimes, Heidelberg
  - Kinderarztpraxis Wirth, Krefeld
  - Studienzentrum Dr. Beate Schwarz, Langenau
  - Dermatologische Praxis Dr. Quist, Mainz
  - Universitätsmedizin Mainz, Zentrum für Kinder- und Jugendmedizin, Mainz
  - Praxis Dr. Panzer, Mannheim
  - Hautarztpraxis Burgstrasse, München
  - Klinikum der Universität München, München
  - Kinderpneumologische Praxis Dr. Funck, Neuss
  - Kinderärztliche Gemeinschaftspraxis Bedikian und Bouikidis, Oberhausen
  - Kinderarztpraxis Dres. Med. Sören Westerholt & Jan Matyas, Wolfsburg
- Netherlands (2):
  - Erasmus MC University Department of Dermatology, Rotterdam
  - St. Franciscus Gasthuis & Vlietland Kindergeneeskunde, Rotterdam
- Poland (3):
  - Dermoklinika Centrum Medyczne, Lodz
  - Dermedic Jacek Zdybski, Ostrowiec Świętokrzyski
  - Kliniczny Szpital Woiewodzki, Rzeszów

IPD SHARING:
Plan to Share IPD: No